CLINICAL TRIAL: NCT03277053
Title: A Mobile Device App to Improve Adherence to an Enhanced Recovery Program for Colorectal Surgery: A Randomized Control Trial
Brief Title: A Mobile Device App to Improve Adherence to an Enhanced Recovery Program for Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Liane S. Feldman (Other)
Collaborators: Society of American Gastrointestinal and Endoscopic Surgeons (Other)
Responsible Party: Sponsor-Investigator, Dr. Liane S. Feldman, Professor, Department of Surgery, McGill University Director, General Surgery Clinical Teaching Unit, Montreal General Hospital. Director, Division of General Surgery at the MUHC and McGill University. Program Director, MIS Fellowship Program., McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: McgillGensurgAPPRCT
Record Dates: First submitted 2017-07-11; First posted 2017-09-08 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Disorders
Keywords: colorectal; laparoscopic; application; ERP; adherence; mobile

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Sham Comparator): Patients receive an ipad with no app.
  Interventions: Other: Control.
- Mobile application no stoma (Experimental): Patients who did not receive a stoma receive an ipad containing the app and are instructed how to use it.
  Interventions: Device: Mobile application
- Mobile application stoma (Experimental): Patients who receive a stoma receive an ipad containing the app and are instructed how to use it.
  Interventions: Device: Mobile application

INTERVENTIONS:
Device: Mobile application — A mobile application designed specifically for colorectal patients treated within an enhanced recovery pathway. Contains information, guidelines, questionnaires and feedback
  Arms: Mobile application no stoma; Mobile application stoma
Other: Control. — Patient receive an ipad with no application.
  Arms: control

SUMMARY:
A randomized control trial on patients undergoing laparoscopic colorectal resection in an Enhanced Recovery Program (ERP). The intervention is delivered via an electronic application containing guidelines, information, and tailored feedback. The hypothesis is that the application will improve adherence to the ERP.

DETAILED DESCRIPTION:
Introduction: Enhanced Recovery Programs (ERP) in colorectal surgery reduce postoperative morbidity and shorten length of hospital stay with no increase in readmission rates. However, poor adherence to ERP elements remains a challenge. Recent studies suggest that the use of mobile device applications has the potential to improve patient compliance with treatment guidelines. We recently developed and pilot tested a mobile app to support an ERP for colorectal surgery which collects patient-reported recovery information and engages patients as stakeholders in their recovery process. The overall aim of this study is to estimate the extent to which the use of this mobile device app impacts adherence to postoperative ERP elements in comparison to standard preoperative education.

Methods. The proposal is for a two-group, assessor-blind, randomized trial including adult patients with colorectal diseases planned for surgical resection.

Participants will be randomly assigned into one of two groups:

1. usual perioperative education and audit, or
2. a mobile device application for postoperative education and self-audit.

The intervention will be delivered through a tablet present at the bedside with an application which links education, recovery planning, and daily self-assessment to a plan of care. It educates patients about daily recovery milestones and track their adherence. The primary outcome will be patient adherence to postoperative enhanced recovery elements. Other targeted outcomes include self-reported recovery, satisfaction and patient activation. According to an a priori power analysis, a sample of 104 patients (52 per group) is targeted for this trial.

Significance: This study will contribute evidence regarding the use of mobile device technology for education and the direct involvement of patients as stakeholders in postoperative recovery.

The study findings have the potential to increase patient engagement in the care pathway, which has the potential to increase compliance to pathway elements and improve postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic colorectal resection.
* Proficient in english or french

Exclusion Criteria:

* intellectual disabilities
* major simultaneous procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Completion of 5 patient-dependent pathway interventions that involve patient participation on the initial 48 hrs after surgery. | postoperative day 2
  Questionnaire including 5 pathway interventions that involve patient participation during the first 48 hours after surgery (mobilization, gum chewing, consumption of oral liquids, breathing exercises, nutritional supplement).

SECONDARY OUTCOMES:
Length of stay | one month
  Number of days spent in the hospital after surgery
Complications | one month
  Comprehensive complication index (CCI)
Successful Recovery | postoperative day 4
  Discharge by postoperative day 4 with no complications.

CONTACTS AND LOCATIONS:
Overall Officials: Liane Feldman, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal general Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No